CLINICAL TRIAL: NCT03524248
Title: Development of Real-time Image-guided Radiotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Camera for study is being repaired
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-6006
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer; Lung Cancer; Skin Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Skin Neoplasms | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: Image guided radiation therapy — Real-time 4D video imaging guidance with combination use of cone-beam computerized tomography (CBCT) useful for daily setup and target motion tracking in advanced image-guided radiotherapy (IGRT).

SUMMARY:
The goal is to achieve the maximal radiotherapy tumor dose while sparing the health tissue and critical structures. On-board cone-beam CT (CBCT) scans are routinely acquired prior to dose delivery and matched with simulation CT at the planned treatment positions. Thus, setup or motion errors can be detected and corrected. However, CBCT is not available for situations with gantry collisions such as WBI and TSEB. More importantly, CBCT cannot reveal any irregular respiration or body movement during beam-on time. Thus, it is essential to develop a real-time image system that can detect organ/body motion during beam-on time, and correlate simulation-planning images with prior treatment CBCT images.In this proposed clinical trial, we will cooperate with a 3D camera company (Xigen LLC) to develop novel 4D video imaging techniques and validate the feasibility and accuracy of 4D video image guidance in correlation with 4D CT/CBCT useful for advanced IGRT.

ELIGIBILITY:
Inclusion Criteria:

* All patients benefit from advanced IGRT can participate to the study except for those emergent and pediatric patients (age <18 years) who require special care or there is no time for the setup the 4D video systems
* The patient population would be selected according to the technical progress and clinical needs

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2012-05-17 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
Develop real-time 4D video imaging guidance with combination use of cone-beam computerized tomography (CBCT) useful for daily setup and target motion tracking in advanced image-guided radiotherapy (IGRT). | 12 years
  Real time 4-D video imaging in combination with CBCT to detect appropriate delivery of radiotherapy

SECONDARY OUTCOMES:
To correlate real-time 4D surface images with the internal structures shown in daily XVI volumetric images | 12 years
  Align 4D surface images with internal structures

OTHER OUTCOMES:
To synchronize the 4D CBCT with real-time stereovisions that would allow us to track any irregular respiration motion useful for gated or target tracked radiotherapy | 12 years
  Synchronization of 4D CBCT with real time stereovision
To validate accuracy and precision of the patient position in special procedures such as stereotactic body radiotherapy (SBRT), total skin electron beam therapy (TSEB), IMRT of H&N cancer, and whole-breast irradiation (WBI) under breast holding | 12 years
  Validation
To determine delivery dose distribution by correlating real-time surface images with the planning volumetric images and dose distribution for radiotherapy | 12 years
  Determine delivery dose distribution at the site or radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States